CLINICAL TRIAL: NCT02751489
Title: Human Phototoxicity Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 18600
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bain De Soliel - Solid (Experimental): All subjects are patched with the same product
  Interventions: Other: Bain De Soliel - Solid

INTERVENTIONS:
Other: Bain De Soliel - Solid — 0.05 gm/cm2 of each test product is applied to duplicate skin sites (approximately 2 x 2 cm each) on the lower or mid-back. After the test articles have dried for 5 to 15 min, the sites are covered by the appropriate patch.

SUMMARY:
To determine the phototoxic potential of a topically applied article in human subjects

ELIGIBILITY:
Inclusion Criteria:

* Be male or female between the ages of 18 and 60 inclusive;
* Be lightly pigmented (Fitzpatrick Skin Type I, II, III);
* Have read and signed the written Informed Consent Form and have completed a Health Insurance Portability and Accountability (HIPAA) Authorization Form in conformance with 45CFR Parts 160 and 164;
* Be in general good health as determined by the subject's medical history and in the discretion of the investigator;

Exclusion Criteria:

* Have a visible sunburn;
* Have a history of sun hypersensitivity/photosensitivity or photosensitive dermatoses;
* Must not have a known sensitivity or allergy against any of the active and non-active ingredients of the test product.
* Have a history of allergies or sensitivities to cosmetics, toiletries or any dermatological products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Intensity of skin reactions is evaluated by 5 point scale | Up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Piscataway, New Jersey, United States